CLINICAL TRIAL: NCT04333875
Title: Morbidity and Mortality Due to Deferral of Aortic Valve Replacement in Patients With Severe Aortic Stenosis - a Collateral Effect of the SARS-CoV-2 Pandemic (AS DEFER)
Brief Title: Morbidity and Mortality Due to Deferral of Aortic Valve Replacement in Patients With Severe Aortic Stenosis
Acronym: AS DEFER
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-00672
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TAVR/SAVR: Patients with critical aortic stenosis as defined by an AVA <0.6 cm2 or a transvalvular mean gradient of >60 mmHg or a history of cardiac decompensation during the previous 3 months or clinical symptoms on minimal exertion (NYHA III) will be allocated to transcatheter aortic valve replacement or surgical aortic valve replacement.
  Interventions: Device: TAVR or SAVR
- Deferred Intervention: Patients with severe but not critical aortic Stenosis will undergo deferred intervention.

INTERVENTIONS:
Device: TAVR or SAVR — Patients with critical aortic stenosis as defined by an AVA <0.6 cm2 or a transvalvular mean gradient of >60 mmHg or a history of cardiac decompensation during the previous 3 months or clinical symptoms on minimal exertion (NYHA III) will be allocated to TAVR or SAVR.
  Groups: TAVR/SAVR

SUMMARY:
Background and Project Rationale:

Degenerative aortic valve stenosis affects 2% of the elderly population aged 70 years or older and progresses insidiously with advancing age [1] before manifesting with symptoms such as decreased exercise tolerance, shortness of breath, chest pain and syncope on exertion. Without aortic valve replacement, the survival prognosis of patients with symptomatic aortic stenosis is poor. In the PARTNER 1B trial, all-cause mortality among 179 inoperable patients with severe symptomatic aortic stenosis allocated to conservative management amounted to 51% at one year [2]. Consistently, prospective registry data reported a mortality rate of 55% at 1 year in 78 patients with severe aortic stenosis undergoing conservative management [3].

The rapid spread of the SARS-CoV-2 pandemic represents an unprecedented challenge for healthcare systems. A limited number of ventilators and ICU beds call for a careful allocation of healthcare resources. On March 20 2020, the Federal Council prohibited elective interventions in all hospitals in Switzerland. Patients with untreated severe aortic stenosis are particularly vulnerable to SARS-CoV-2 infection [4] and face the dual risk of cardiac death from aortic stenosis on one side, and death from acute respiratory distress syndrome secondary to SARS-CoV-2 infection on the other. While the balance between the two risks is a matter of clinical judgement, the investigators established an algorithm for the management of patients with severe aortic stenosis during the SARS-CoV-2 pandemic. Patients with aortic stenosis deemed critical will undergo valvular replacement in spite of the ongoing pandemic while patients with severe but not critical aortic stenosis will undergo deferred intervention once the number of new SARS-CoV-2 infections flattens.

In the current situation, aortic valve replacement in patients with severe, non-critical aortic stenosis will be deferred in order to give priority to SARS-CoV-2 patients. This unique situation allows the investigators to study the effect of deferral of aortic valve replacement in patients with severe aortic stenosis.

The study is an amendment to the Swiss-TAVI registry. In contrast to the Swiss-TAVI registry, patients are not enrolled at the time of aortic valve replacement, but already at the time of referral for aortic valve replacement.

Primary Objective:

The aim of the present observational study is to explore the effect of deferral of valvular replacement in patients with severe but not critical aortic stenosis on morbidity and mortality. The primary objective is to describe rates of morbidity and mortality among patients with severe but not critical aortic stenosis in the interval from referral/indication for valvular replacement to intervention.

Project Design:

The study is a prospective cohort study of patients with severe aortic stenosis referred for aortic valve replacement. All referrals for aortic valve replacement will be allocated to either "transcatheter aortic valve replacement (TAVR)/ surgical aortic valve replacement (SAVR) (standard of care)" or "deferred intervention" based on prespecified criteria. Patients with critical aortic stenosis as defined by an aortic valve area (AVA) <0.6 cm2 or a transvalvular mean gradient of >60 mmHg or a history of cardiac decompensation during the previous 3 months or clinical symptoms on minimal exertion (NYHA III) will be allocated to TAVR or SAVR. All other patients with severe aortic stenosis defined by an AVA <1.0 cm2 will be scheduled for a deferred intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients with severe AS defined by an AVA <1cm2 or AVA indexed to BSA of <0.6 cm2/m2, including low-flow severe aortic stenosis defined by SVI <35ml/m2.

Exclusion Criteria:

* Life expectancy <1 year irrespective of severe AS.
* Severe dementia defined as MMS-Test <16 points.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The project population comprises all consecutive patients with severe aortic stenosis referred for aortic valve replacement (TAVR or SAVR) since March 20 2020 until the end of the prohibition of elective interventions in Switzerland.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Composite of all-cause mortality, disabling and non-disabling stroke, and hospitalization for heart failure | Assessed at 6 months after indication/referral for aortic valve replacement.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Pilgrim, MD, Principal Investigator — University of Bern, Switzerland
Locations (1):
- Department of Cardiology, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Yadgir S, Johnson CO, Aboyans V, Adebayo OM, Adedoyin RA, Afarideh M, Alahdab F, Alashi A, Alipour V, Arabloo J, Azari S, Barthelemy CM, Benziger CP, Berman AE, Bijani A, Carrero JJ, Carvalho F, Daryani A, Duraes AR, Esteghamati A, Farid TA, Farzadfar F, Fernandes E, Filip I, Gad MM, Hamidi S, Hay SI, Ilesanmi OS, Naghibi Irvani SS, Jurisson M, Kasaeian A, Kengne AP, Khan AR, Kisa A, Kisa S, Kolte D, Manafi N, Manafi A, Mensah GA, Mirrakhimov EM, Mohammad Y, Mokdad AH, Negoi RI, Thi Nguyen HL, Nguyen TH, Nixon MR, Otto CM, Patel S, Pilgrim T, Radfar A, Rawaf DL, Rawaf S, Rawasia WF, Rezapour A, Roever L, Saad AM, Saadatagah S, Senthilkumaran S, Sliwa K, Tesfay BE, Tran BX, Ullah I, Vaduganathan M, Vasankari TJ, Wolfe CDA, Yonemoto N, Roth GA; Global Burden of Disease Study 2017 Nonrheumatic Valve Disease Collaborators. Global, Regional, and National Burden of Calcific Aortic Valve and Degenerative Mitral Valve Diseases, 1990-2017. Circulation. 2020 May 26;141(21):1670-1680. doi: 10.1161/CIRCULATIONAHA.119.043391. Epub 2020 Mar 29. PMID 32223336
- [Result] Leon MB, Smith CR, Mack M, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Brown DL, Block PC, Guyton RA, Pichard AD, Bavaria JE, Herrmann HC, Douglas PS, Petersen JL, Akin JJ, Anderson WN, Wang D, Pocock S; PARTNER Trial Investigators. Transcatheter aortic-valve implantation for aortic stenosis in patients who cannot undergo surgery. N Engl J Med. 2010 Oct 21;363(17):1597-607. doi: 10.1056/NEJMoa1008232. Epub 2010 Sep 22. PMID 20961243
- [Result] Wenaweser P, Pilgrim T, Kadner A, Huber C, Stortecky S, Buellesfeld L, Khattab AA, Meuli F, Roth N, Eberle B, Erdos G, Brinks H, Kalesan B, Meier B, Juni P, Carrel T, Windecker S. Clinical outcomes of patients with severe aortic stenosis at increased surgical risk according to treatment modality. J Am Coll Cardiol. 2011 Nov 15;58(21):2151-62. doi: 10.1016/j.jacc.2011.05.063. PMID 22078420
- [Result] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076